CLINICAL TRIAL: NCT03570788
Title: Health-related Quality of Life Among Patients Amputated Due to Peripheral Arterial Disease
Brief Title: HRQoL Among Patients Amputated Due to Peripheral Arterial Disease
Status: Completed | Type: Observational
Sponsor: Jonas Malmstedt (Other)
Responsible Party: Sponsor-Investigator, Jonas Malmstedt, Co - Principal Investigator, M.D Ph.D., Karolinska Institutet
Organization: Karolinska Institutet (Other)
Other Study IDs: 2014/801-31/1
Record Dates: First submitted 2018-06-13; First posted 2018-06-27 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Quality of Life; Amputation; Peripheral Arterial Disease; Prosthesis User
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Amputation, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Amputation — Major amputation defined as at or above ankle

SUMMARY:
A prospective cohort study over the prosthetic use among patients amputated after vascular disease and the impact of their HRQoL.

ELIGIBILITY:
Inclusion Criteria:

* Patients amputated at femoral, knee or tibial level due to peripheral arterial disease

Exclusion Criteria:

* Patients not able to provide informed consent
* Patients not able to verbally express their experience of the amputation.
* Patients that not speak Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients amputated at Södersjukhuset during 2014-2018 are reviewed based on criteria for inclusion and exclusion. All patients that meets the inclusion criteria during the period will be contacted by the researcher in connection with the amputation and informed about the study.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2014-09-12 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Change in Health related quality of life according to EQ-5D | 1 year
  The change in HRQoL between baseline and after 1 year. Measured with EQ-5D-3L

SECONDARY OUTCOMES:
Proportion of patients using prosthesis | 1 year after the amputation
  Prosthesis use after a major amputation is measured with Stanmore mobility grade

CONTACTS AND LOCATIONS:
Overall Officials: Eva Torbjörnsson, Principal Investigator — Department of Clinical Science and Education, Södersjukhuset, Karolinska Institutet
Locations (1):
- Department of Clinical Science and Education, Södersjukhuset, Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No